CLINICAL TRIAL: NCT01426893
Title: Observational Study to Evaluate the Correctness of the Use of Inhaler Device in Patients With Asthma or Chronic Obstruct
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RRS-XXX-2011/1
Record Dates: First submitted 2011-08-29; First posted 2011-09-01 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Asthma,; Chronic Obstructive Pulmonary Disease
Keywords: Respiratory disease; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Respiration Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: The inhaler device usage in patients with asthma or COPD

SUMMARY:
The correct use of inhalation devices is an inclusion criterion for all studies comparing inhaled treatments. In real life, however, patients may make many errors with their usual inhalation device, which may negate the benefits observed in clinical trials. In real life, many errors seem to be made, but no wide-scale evaluation has been performed. The correct use of inhalation devices is essential to ensure the effectiveness of the treatment. It has been recently demonstrated that inhaler misuse is associated with decreased asthma control in asthmatics treated with an inhaled corticosteroid. The aim of our observational study was to evaluate the inhaler device usage in patients with asthma or chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Observational study to evaluate the correctness of the use of inhaler device in patients with asthma or chronic obstruct

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent
* Females or males aged > 18 years

Exclusion Criteria:

- If participating in any other clinical trial, the subject cannot take part in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Speciality care clinics
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Investigator's evaluation of the correctness of patients' usage of inhaler device in patients with asthma or COPD assesses by investigator/pulmonologist | 12 weeks

SECONDARY OUTCOMES:
Global assessment of disease control, done by investigator. Investigator will globally assess the disease control by one on three categories: 'fully controlled', 'partially controlled', 'uncontrolled'. | 12 weeks
Evaluation of patients' perception of the inhaler device and their perspective of symptom control and impact on daily life, by using the patient's questionnaire | 12 weeks
Evaluation of the influence of practical education of the patients (performed by physician and/or nursing staff) on all above parameters/assessments | 12 weeks
Collection of local demographics data in patients with asthma or COPD | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Predrag Rebic, Prof.dr, Principal Investigator — Clinical Center of Serbia, Belgrade
Locations (5):
- Serbia (5):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Sombor